CLINICAL TRIAL: NCT00873275
Title: Phase I Study of Ursodeoxycholic Acid (Ursodiol)in Combination With 5-Fluorouracil, Leucovorin, Oxaliplatin and Bevacizumab in Patients With Metastatic Colorectal Cancer
Brief Title: Ursodiol, Combination Chemotherapy, and Bevacizumab in Treating Patients With Stage IV Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08005; P30CA033572 (NIH); CHNMC-08005; CDR0000637521 (Registry Identifier: NCI PDQ); NCI-2010-00926 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin; Ursodeoxycholic Acid; Gene Expression Profiling; Polymerase Chain Reaction; Blotting, Western; Immunohistochemistry; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ursodiol, combination chemotherapy, bevacizumab) (Experimental): Patients receive oral ursodiol twice daily on days 1-28 (days -6 to 28 of course 1), leucovorin calcium IV over 2 hours on days 1 and 15, fluorouracil IV over 46 hours on days 1-2 and 15-16, and oxaliplatin IV over 2 hours and bevacizumab IV over 30-90 minutes on days 1 and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: FOLFOX regimen; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Drug: ursodiol; Genetic: RNA analysis; Genetic: gene expression analysis; Genetic: polymerase chain reaction; Genetic: western blotting; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: positron emission tomography (PET)

INTERVENTIONS:
Biological: bevacizumab — 5mg/kg IV day 1 and 15 of each 28 day course of treatment
Drug: FOLFOX regimen — Leucovorin, 5-FU and Oxaliplatin
Drug: fluorouracil — 400 mg/m2 IV bolus immediately following leucovorin on days 1 and 15 of a 28 day course of treatment. Then 2.4 gm/m2 IV continuous infusion over 46 hours immediately following bolus dose on days 1 and 2 and 15 and 16 of a 28 day course of treatment
Drug: leucovorin calcium — 400 mg/m2 IV infusion over 2 hours on days 1 and 15 of a 28 day course of treatment.
Drug: oxaliplatin — 85 mg/m2 IV infusion over 2 hours on days 1 and 15 of a 28 day course of treatment.
Drug: ursodiol — Dose escalation in cohorts (3 patients/cohort) from an initial dose of 125 mg PO BID through 625 mgs PO BID beginning on Day -6 from infusion of bevacizumab and FOLFOX continuing for the duration of the treatment.
Genetic: RNA analysis — Analysis on discard tissues
Genetic: gene expression analysis — Determined in normal and malignant tissues in patients who undergo surgical resection after treatment on this trial
Genetic: polymerase chain reaction — Analysis on discard tissues
Genetic: western blotting — Determined on blood collected at Day -6, Day 0 and Day 7 (1 week after the first cycle of chemotherapy) from treatment and at the end of treatment
Other: immunohistochemistry staining method — Performed on tumor blocks from the primary and the metastases from the patients on study
Other: laboratory biomarker analysis — Performed on blood collected at Day -6, Day 0 and Day 7 (1 week after the first cycle of chemotherapy) from treatment and at the end of treatment
Other: pharmacological study — Day 0, day 7 before treatment, 1/2 hour after the start of treatment, 1, 2, 3, 4, and 8 hours after the start of treatment.
Procedure: positron emission tomography (PET) — Patients will undergo PET scan imaging as part of their original staging or at baseline. If the PET scan was more than 2 weeks prior to Day 0 from study treatment, there will be a PET scan at Day 0. In any case there will be a PET scan when the patient completes treatment.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ursodiol, oxaliplatin, leucovorin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of colorectal cancer by blocking blood flow to the tumor. Giving ursodiol together with leucovorin calcium, fluorouracil, oxaliplatin, and bevacizumab may be an effective treatment for colorectal cancer.

PURPOSE: This phase I trial is studying the side effects and best dose of ursodiol when given together with combination chemotherapy and bevacizumab in treating patients with stage IV colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the active dose and/or maximum tolerated dose of ursodiol when given in combination with fluorouracil, leucovorin calcium, oxaliplatin (FOLFOX regimen), and bevacizumab in patients with metastatic colorectal cancer.
* To determine the pharmacokinetics of ursodiol when given with this regimen.

Secondary

* To determine the systemic metabolic effects of ursodiol activation of nuclear receptor farnesoid X receptor (FXR) in glucose and lipid metabolism.
* To develop assays to detect ursodiol activation of FXR.
* To identify and evaluate potential serum biomarkers of FXR activation.
* To determine genes regulated by activation of FXR at target tissues.

OUTLINE: This is a dose-escalation study of ursodiol.

Patients receive oral ursodiol twice daily on days 1-28 (days -6 to 28 of course 1), leucovorin calcium intravenously (IV) over 2 hours on days 1 and 15, fluorouracil IV over 46 hours on days 1-2 and 15-16, and oxaliplatin IV over 2 hours and bevacizumab IV over 30-90 minutes on days 1 and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Blood sample is collected periodically for pharmacokinetic studies. Samples are also analyzed for the role of nuclear receptor farnesoid X receptor (FXR) in glucose uptake and metabolism using PET scan imaging, an oral glucose tolerance test, and HbA1c levels; the effects of FXR activation on lipid metabolism; and a marker for response to FXR activation via western blot. Available formalin-fixed paraffin-embedded tumor tissue blocks are analyzed for FXR expressing via IHC; expression of known FXR target genes via RNA analysis and real-time PCR; and expression of genes involved in glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced, biopsy proven metastatic colorectal cancer
* Karnofsky Performance Status >= 80
* Prior therapy completed at least 3 weeks before protocol treatment initiation with recovery from any side-effects
* Serum albumin and prealbumin within normal limits
* Alanine aminotransferase (ALT) within 3 x upper limit of normal
* Alkaline phosphatase within 3 x upper limit of normal
* Serum bilirubin within normal limits
* Absolute neutrophil count >= 1500/ul
* Serum creatinine within 1.5 x upper limit of normal
* Ability to understand and sign an institutional review board (IRB) approved informed consent
* Ability to use appropriate contraception and no evidence of pregnancy in female patients of reproductive potential

Exclusion Criteria:

* Significant medical or psychiatric condition that would make treatment unsafe
* Use of systemic steroids use within 7 days from start of trial
* Nursing women
* Patients unable to comply with protocol related studies and follow up
* Weight loss of greater than 10% in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-03-11 (Actual); Primary Completion 2012-09-25 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose of ursodiol | 28 days from the start of treatment
Toxicities as assessed by NCI CTCAE 3.0 | 28 days after the last cycle of treatment
Survival | 2 years after treatment
Time to failure | 2 years after treatment
Pharmacokinetics of ursodiol | 8 days after start of treatment during course 1

CONTACTS AND LOCATIONS:
Overall Officials: Lily L. Lai, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States